CLINICAL TRIAL: NCT04170855
Title: Evaluation of Kidney Medullary Sodium Content Using 23Na MRI to Understand and Predict Diuretic Resistance
Brief Title: Kidney Sodium Content in Cardiorenal Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Chris McIntyre, Professor of Medicine, Medical Biophysics and Pediatrics, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 114884
Record Dates: First submitted 2019-10-21; First posted 2019-11-20 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Cardio-Renal Syndrome
Keywords: kidney sodium content; Sodium MRI
MeSH Terms: conditions — Cardio-Renal Syndrome | interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Furosemide Injection (Other): Patients with diuretic resistance:
  The presence of diuretic resistance, defined as having clinical signs of fluid overload despite diuretic therapy (this information is routinely collected at each clinical visit). "Fluid overload" is defined as the presence of at least two of the following clinical features:
  * Peripheral or sacral oedema
  * Jugular venous distension ≥ 7 cm
  * Radiographic pulmonary oedema or pleural effusion
  * Enlarged liver or ascites
  * Pulmonary rales, paroxysmal nocturnal dyspnoea, or orthopnoea
  * Point of Care UltraSound (POCUS) evidence of congestion. Inferior Vena Cava diameter >2.5 cm and/or failure to collapse at least 50% with sharp inspiration
  Interventions: Drug: Furosemide Injection

INTERVENTIONS:
Drug: Furosemide Injection — We will measure kidney sodium content in patient with cardiorenal syndrome. we will inject within the week of this first measurement furosemide only in patient who will be resistant to diuretics (Based on these parameters, diuretic response will be defined as:
  * A reduction in fractional spot urinary sodium
  * An increase in urinary volume
  * A >1 kg reduction in body weight within 24 hours from diuretic administration (extrapolation of guidance on management of acute HF) and we will do another measurement of kidney sodium content after furosemide injection.

SUMMARY:
Diuretic therapy is the cornerstone of the management of fluid overload in heart failure. Resistance to diuretic therapy is the most common reason for treatment failure in patients affected by the combination of heart failure and kidney disease. Currently, there is no way of predicting whether heart failure patients will develop resistance to diuretic therapy and what dose of diuretic is necessary to overcome diuretic resistance. Answering these questions would allow doctors to be able to prescribe an accurate dose of diuretic therapy to prevent diuretic resistance and potential side effects of an excessive diuretic dose.

With magnetic resonance imaging, it is possible to measure the kidney sodium (salt) content and observe the diuretic response in patients with heart failure and kidney disease. The investigators speculate that measuring kidney sodium content will allow to predict diuretic response in these patients.

The aim of this study is to compare the kidney sodium content in patients with chronic cardiorenal syndrome with and without diuretic resistance. Secondly, in a sample of patients with diagnosed diuretic resistance,the aim will be to observe the changes in kidney sodium content induced by an additional dose of diuretic therapy and to observe whether these changes are associated with a response to diuretic therapy.

DETAILED DESCRIPTION:
This is a prospective, interventional, pilot study involving patients recruited from the Heart Failure outpatient clinic at St. Joseph's Hospital in London, Ontario. Depending on scanner availability, the study visits may also take place at Robarts Research Institute, University of Western Ontario. All eligible patients who consent to take part in the study will undergo one study visit. During this visit, all study participants will undergo a combined proton (1H) and 23Na MRI scan of their kidneys to measure kidney sodium content. Prior to the scan, all participants will be asked to complete a questionnaire, will have their fluid volume measured using bioimpedance spectroscopy, will have their heart failure classified using the NYHA system, will have their weight taken using a clinical scale, and will have their sitting blood pressure and heart rate measured three times consecutively using a standard automatic blood pressure monitor. In addition to this, all participants will undergo a research focused echocardiogram, provide a spot urine sample and have blood work collected. All participants will be responsible to complete a 24-hour urine volume test the day before the study visit and bring the special container to the team on the visit day.

Study participants who meet the criteria for diuretic resistance will undergo a second study visit within one week of the first one. During this visit, participants will receive an additional intravenous dose of diuretic (furosemide) and they will subsequently undergo a second proton and 23Na MRI scan of their kidneys. Prior to the scan participants will undergo the same study procedures as in visit one excluding the questionnaire. In addition to this, participants will be responsible to record their weight at home the morning before the visit and bring their weight to the study team. After the scan, all participants will have their blood pressure, heart, rate, and weight measured again, and will be asked to complete a 24-hour urine collection. Furthermore, participants will be asked to take their weight using a home scale the morning after the scan and a member of the research team will phone the participants to collect this information.

ELIGIBILITY:
Inclusion Criteria for Visit 1

* Clinico-pathological diagnosis of heart failure
* Age ≥ 18 years
* Estimated GFR ≥ 15 mL/min/1.73m2
* Receiving loop diuretics for at least a week at ≥ 40 mg/day (furosemide) or 2 mg/day (bumetanide), either orally or intravenously
* Willing and able to provide consent

Inclusion Criteria for Visit 2 · Patients from visit 1 with diuretic resistance

Exclusion Criteria for Visit 1 Direct contraindications to MR scanning (implanted materials etc.)

* Additional diuretic types other than spironolactone/epleronone/metolazone/finerenone
* Liver disease with hepato-renal syndrome
* Pregnant, breastfeeding or intending pregnancy
* Kidney malformation leading to chronic kidney disease (for example polycystic kidney)
* Unable to provide consent

Exclusion criteria for Visit 2

· Hypokalemia (serum potassium <3.5 mmol/l)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Medullary sodium concentration | Through MRI, an average of 60 minutes
  To demonstrate a statistically significant difference in medullary sodium concentration of at least 100 mmol/L between patients with chronic cardiorenal syndrome who are responsive versus patients who are resistant to their current diuretic therapy.

SECONDARY OUTCOMES:
Corticomedullary sodium gradient | Through MRI, an average of 60 minutes
  To demonstrate a difference in corticomedullary sodium gradient between patients with chronic cardiorenal syndrome who are responsive versus patients who are resistant to their current diuretic therapy.
Change in medullary sodium concentration | Through MRI, an average of 60 minutes
  To demonstrate a change in medullary sodium concentration compared to baseline in patients with chronic cardiorenal syndrome and diuretic resistance who show a clinical response to an additional diuretic dose, assessed by the lost of weight.
Change in corticomedullary sodium gradient | Through MRI, an average of 60 minutes
  To demonstrate a change in corticomedullary sodium gradient compared to baseline in patients with chronic cardiorenal syndrome and diuretic resistance who show a clinical response to an additional diuretic dose
Correlation between kidney sodium content and renal function | Through one study visit, and average of 3 hours
  To investigate the correlation between kidney sodium content and renal function assessed by GFR measurement (mL/min/1.73m2)
Correlation between kidney sodium content and biological cardiac biomarker | Through one study visit, and average of 3 hours
  To investigate the correlation between kidney sodium content and cardiac biomarkers assessed by NT-ProBNP
Correlation between kidney sodium content and inflammation | Through one study visit, and average of 3 hours
  To investigate the correlation between kidney sodium content and inflammation biomarkers assessed by CRP (mg/dL)
Correlation between kidney sodium content and NYHA | Through one study visit, an average of 3 hours
  To investigate the correlation between kidney sodium content and NYHA class (no unit, scale from 0 to 4)
Correlation between kidney sodium content and echocardiography | Through one study visit, an average of 3 hours
  To investigate the correlation between kidney sodium content and left ejection fraction (in %)
Correlation between kidney sodium content and Bioimpedance spectroscopy | Through one study visit, an average of 3 hours
  To investigate the correlation between kidney sodium content and extra cellular volume content (in liters) measured by bioimpedance spectroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher W McIntyre, MD, Principal Investigator — Western University
Locations (1):
- Heart Failure Clinic | St. Joseph's Health Care London, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mosterd A, Hoes AW. Clinical epidemiology of heart failure. Heart. 2007 Sep;93(9):1137-46. doi: 10.1136/hrt.2003.025270. PMID 17699180
- [Background] Chioncel O, Mebazaa A, Harjola VP, Coats AJ, Piepoli MF, Crespo-Leiro MG, Laroche C, Seferovic PM, Anker SD, Ferrari R, Ruschitzka F, Lopez-Fernandez S, Miani D, Filippatos G, Maggioni AP; ESC Heart Failure Long-Term Registry Investigators. Clinical phenotypes and outcome of patients hospitalized for acute heart failure: the ESC Heart Failure Long-Term Registry. Eur J Heart Fail. 2017 Oct;19(10):1242-1254. doi: 10.1002/ejhf.890. Epub 2017 Apr 30. PMID 28463462
- [Background] McCullough PA, Kellum JA, Haase M, Muller C, Damman K, Murray PT, Cruz D, House AA, Schmidt-Ott KM, Vescovo G, Bagshaw SM, Hoste EA, Briguori C, Braam B, Chawla LS, Costanzo MR, Tumlin JA, Herzog CA, Mehta RL, Rabb H, Shaw AD, Singbartl K, Ronco C. Pathophysiology of the cardiorenal syndromes: executive summary from the eleventh consensus conference of the Acute Dialysis Quality Initiative (ADQI). Contrib Nephrol. 2013;182:82-98. doi: 10.1159/000349966. Epub 2013 May 13. PMID 23689657
- [Background] Clark AL, Kalra PR, Petrie MC, Mark PB, Tomlinson LA, Tomson CR. Change in renal function associated with drug treatment in heart failure: national guidance. Heart. 2019 Jun;105(12):904-910. doi: 10.1136/heartjnl-2018-314158. PMID 31118203
- [Background] Jamison RL. The renal concentrating mechanism: micropuncture studies of the renal medulla. Fed Proc. 1983 May 15;42(8):2392-7. PMID 6341087
- [Background] Faris RF, Flather M, Purcell H, Poole-Wilson PA, Coats AJ. Diuretics for heart failure. Cochrane Database Syst Rev. 2012 Feb 15;(2):CD003838. doi: 10.1002/14651858.CD003838.pub3. PMID 22336795
- [Background] Maril N, Rosen Y, Reynolds GH, Ivanishev A, Ngo L, Lenkinski RE. Sodium MRI of the human kidney at 3 Tesla. Magn Reson Med. 2006 Dec;56(6):1229-34. doi: 10.1002/mrm.21031. PMID 17089361
- [Background] Maril N, Margalit R, Mispelter J, Degani H. Sodium magnetic resonance imaging of diuresis: spatial and kinetic response. Magn Reson Med. 2005 Mar;53(3):545-52. doi: 10.1002/mrm.20359. PMID 15723399
- [Derived] Akbari A, Lemoine S, Salerno F, Marcus TL, Duffy T, Scholl TJ, Filler G, House AA, McIntyre CW. Functional Sodium MRI Helps to Measure Corticomedullary Sodium Content in Normal and Diseased Human Kidneys. Radiology. 2022 May;303(2):384-389. doi: 10.1148/radiol.211238. Epub 2022 Feb 8. PMID 35133199